CLINICAL TRIAL: NCT00094952
Title: Biomarkers and Early Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Other Study IDs: IA0054; AG022374
Record Dates: First submitted 2004-10-28; First posted 2004-10-29 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Alzheimer's Disease
Keywords: Mild Cognitive Impairment; Alzheimer's disease; magnetic resonance imaging; cerebrospinal fluid (CSF) biomarkers
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The main goal of this project is to use imaging and biomarkers to identify cognitively normal elderly people who are at increased risk for developing mild cognitive impairment (MCI). MCI is the earliest clinically detectable evidence for brain changes due to Alzheimer's disease (AD). The second goal of this project is to describe the inter-relationships among anatomical biomarkers, cerebrospinal fluid biomarkers, and cognition measures in those elderly people who develop MCI.

DETAILED DESCRIPTION:
The goal of this project is to use magnetic resonance imaging (MRI) and cerebrospinal fluid (CSF) biomarkers to identify cognitively normal participants who show the earliest clinically detectable brain changes of Alzheimer's disease (AD).

The major hypothesis for this study is that CSF P-tau231 measurement improves the accuracy of MRI and cerebrospinal fluid (CSF) measurements in predicting mild cognitive impairment (MCI). Validation of this hypothesis can lead to improved diagnostic tools for detecting AD as early as possible.

This 5-year longitudinal study will involve a baseline exam and two 18-month followup exams. Participants will undergo MRI scans, CSF collection and blood samples, neuropsychological performance testing, and medical, neurological and psychiatric assessment. The screening and diagnostic evaluations will be carried out by the New York University Alzheimer Disease Core Center (ADCC) and the NYU Center for Brain Health.

This study will enroll a minimum of 80 cognitively normal participants, 60 to 80 years of age, with English as their first language, with about 12 years of formal education, and who are living in the metropolitan New York City area. All participants will receive baseline and follow-up evaluations to rule out confounding medical, neurological, and psychiatric conditions that could affect cognition. The study coordinator will maintain 6-month telephone contact with all participants and their caregivers who are part of the project.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of either sex, with a high school education, and between the ages of 60 and 80 years living in the New York City metropolitan area.
* Minimum of 12 years education.
* Participants will be classified as within normal limits on medical, psychiatric and neuropsychological examinations (performance that is better than -1.5 sd of the NYU norm based WMS-R delayed memory index).
* Participants will have a global deterioration scale (GDS)=1 or 2. Those enrolled in the High-Risk group will have a GDS=2 and have a score of >25 on the Memory Complaint Questionnaire (MCQ). In high risk memory loss cases, an informed family member or caregiver will be interviewed to confirm that the participant can perform specific tasks.

Exclusion Criteria:

* Past history or MRI evidence of brain damage including significant trauma, stroke, hydrocephalus, lacunar infarcts, seizures, mental retardation or serious neurological disorder.
* Significant history of alcoholism or drug abuse.
* History of psychiatric illness (e.g., schizophrenia, mania, Post-Traumatic Stress Disorder [PTSD], or depression).
* Any focal neurological signs or significant neuropathology.
* A score of 4 or greater on the Modified Hachinski Ischemia Scale, indicative of cerebrovascular disease.
* A total score of 16 or more on the Hamilton Depression Scale to exclude possible cases of primary depression.
* Evidence of clinically relevant and uncontrolled hypertensive, cardiac, pulmonary, vascular, metabolic or hematologic conditions.
* Physical impairment of such severity as to adversely affect the validity of psychological testing.
* Hostility or refusal to cooperate.
* Any prosthetic devices (e.g., pacemaker or surgical clips) that could be affected by the magnetic field employed during MRI imaging.
* History of familial early onset dementia.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2003-04; Study Completion 2008-03

CONTACTS AND LOCATIONS:
Overall Officials: Mony J. de Leon, Ed.D., Principal Investigator — Center for Brain Health, Silberstein Institute
Locations (1):
- Center for Brain Health, Silberstein Institute, New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Rusinek H, De Santi S, Frid D, Tsui WH, Tarshish CY, Convit A, de Leon MJ. Regional brain atrophy rate predicts future cognitive decline: 6-year longitudinal MR imaging study of normal aging. Radiology. 2003 Dec;229(3):691-6. doi: 10.1148/radiol.2293021299. PMID 14657306
- [Background] Buerger K, Teipel SJ, Zinkowski R, Blennow K, Arai H, Engel R, Hofmann-Kiefer K, McCulloch C, Ptok U, Heun R, Andreasen N, DeBernardis J, Kerkman D, Moeller H, Davies P, Hampel H. CSF tau protein phosphorylated at threonine 231 correlates with cognitive decline in MCI subjects. Neurology. 2002 Aug 27;59(4):627-9. doi: 10.1212/wnl.59.4.627. PMID 12196665
- [Background] de Leon MJ, Segal S, Tarshish CY, DeSanti S, Zinkowski R, Mehta PD, Convit A, Caraos C, Rusinek H, Tsui W, Saint Louis LA, DeBernardis J, Kerkman D, Qadri F, Gary A, Lesbre P, Wisniewski T, Poirier J, Davies P. Longitudinal cerebrospinal fluid tau load increases in mild cognitive impairment. Neurosci Lett. 2002 Nov 29;333(3):183-6. doi: 10.1016/s0304-3940(02)01038-8. PMID 12429378
- See also: Silberstein Institute for Aging and Dementia, New York University School of Medicine — http://aging.med.nyu.edu/